CLINICAL TRIAL: NCT05830032
Title: Impact of Dietary Fibre Consumption on Digestive Comfort
Acronym: Fibrecomf
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Glasgow (Other)
Collaborators: Mondelēz International, Inc. (Industry)
Responsible Party: Principal Investigator, Christine Edwards, Professor, University of Glasgow
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CP/2294514
Record Dates: First submitted 2023-03-24; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Gastrointestinal Discomfort
MeSH Terms: interventions — Inulin; maltodextrin

STUDY DESIGN:
Intervention Model Description: Healthy adults will be recruited for this single blind randomised controlled cross over study. Participants will be provided with powdered fibres and a non-fibre control (blinded) with detailed instruction on how to dilute these to produce an orange flavoured drinks. They will record any digestive symptoms experienced over four different 7-day intervention arms. The participants will record their bowel habits (stool frequency and form) during these intervention periods and provide stool samples before and after each period from which we will measure pH, water content and short chain fatty acids (SCFA) concentration.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Soluble Corn fibre (Experimental): Soluble corn fibre (SCF) (15g fibre/day)
  Interventions: Dietary Supplement: Soluble corn fibre
- Inulin (Experimental): Inulin (In) (15g fibre/day)
  Interventions: Dietary Supplement: Inulin
- Soluble corn fibre and inulin (Experimental): SCF + In (15g/day fibre)
  Interventions: Dietary Supplement: soluble corn fibre and inulin
- Control (Maltodextrin) (Placebo Comparator): Control (Maltodextrin) (0g fibre)
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Soluble corn fibre — As a powdered beverage
  Arms: Soluble Corn fibre
Dietary Supplement: Inulin — As a powdered beverage
  Arms: Inulin
Dietary Supplement: soluble corn fibre and inulin — As a powdered beverage
  Arms: Soluble corn fibre and inulin
Dietary Supplement: Maltodextrin — As a powdered beverage
  Other Names: Placebo
  Arms: Control (Maltodextrin)

SUMMARY:
The purpose of this randomised, placebo-controlled, cross-over study is to compare the impact different fibres have on gastrointestinal symptoms when they are consumed individually or as mixtures in healthy adults. The impact of different fibres on the experience of symptoms and stool parameters will be assessed.

DETAILED DESCRIPTION:
Global sugar consumption is higher than recommended and there are suggestions that this may be linked to the development of non-communicable diseases including dental caries, and obesity. There are many alternatives to sugars that can be used in foods including certain dietary fibres such as inulin or fructo-oligosaccharides. Most dietary fibres can be fully or partially fermented in the colon by the commensal microbiota, producing beneficial bioactive molecules. However, the rapid production of gas during the fermentation of highly soluble fermentable fibres may cause undesirable symptoms for some people. Dietary exposure to the fibres used in food reformulation, including inulin and soluble corn fibre, is increasing and the impact this may have on gastrointestinal symptoms is unclear. The impact of fibres with different physicochemical characteristics and fermentabilities may differ when consumed in mixtures compared to individually.

The aim of this study is to investigate the impact different fibres have on gastrointestinal symptoms when they are consumed individually or as mixtures and how this relates to the composition of the stool.

ELIGIBILITY:
Inclusion criteria:

* Self-reported healthy adults (aged 18-65y)
* Non-smokers

Exclusion criteria:

* Individuals with any allergies or conditions affecting bowel health e.g. inflammatory bowel disease (Crohn's disease or ulcerative colitis), irritable bowel syndrome, coeliac disease or diverticular disease
* Individuals who are pregnant or are trying to get pregnant
* Individuals with any food allergies
* Individuals who have taken antibiotics in the past 3 months
* Individuals who regularly take medication that may modify gastrointestinal function e.g. prokinetic agents (e.g. metoclopramide), antiemetics, constipation treatments (e.g. lactulose, polyethylene glycol)
* Individuals who consume ≥25g fibre per day

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-05-20 (Estimated); Study Completion 2023-10-25 (Estimated)

PRIMARY OUTCOMES:
Symptom frequency and intensity scores | over 7 days
  Symptom frequency and intensity scores for abdominal pain, abdominal bloating and flatulence individually will be reported during each 7-day feeding period. Symptoms will be analysed individually and in combination to create a composite score using a visual analogue scale. This entails making a mark on a horizontal line of 10cm indicating 0 (no symptom) to 10 (worst imaginable symptom). Participants will record the occurrence of each symptom and rate the severity using this scale. The combined score is the sum of each of the symptoms.

SECONDARY OUTCOMES:
Stool frequency | over 7 days
  Diary
Stool form using the Bristol stool chart | Over 7 days
  Diary for each event
Stool water content | Day 1 and day 7
  2 samples each week
Stool acidity | Day 1 and day 7
  2 samples each week
Stool SCFA concentrations | Day 1 and day 7
  2 samples each week

CONTACTS AND LOCATIONS:
Overall Officials: Christine A Edwards, PhD, Principal Investigator — University of Glasgow; Ada L Garcia, PhD, Principal Investigator — University of Glasgow
Locations (1):
- Human Nutrition New Lister Building, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No